CLINICAL TRIAL: NCT03569202
Title: A Randomized, Active-controlled, Parallel, Double-blind Study on the Safety, Ocular Tolerability and Efficacy of Piiloset Trehalose Emulsion Eye Drop in Adult Patients With Moderate or Severe Dry Eye
Brief Title: Piiloset Trehalose Emulsion Eye Drop Study in Moderate or Severe Dry Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: Finnsusp Ltd. (Industry); 4Pharma Ltd. (Industry); Business Finland (Other)
Responsible Party: Principal Investigator, Kai Kaarniranta, MD, PhD, Professor, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5503762
Record Dates: First submitted 2018-04-24; First posted 2018-06-26 (Actual); Results first posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-11

CONDITIONS: Dry Eye Syndrome
Keywords: Lubricant Eye Drops; Moderate or Severe Dry Eye; Hyaluronic Acid; Trehalose; Disaccharides; Polysaccharides; Fatty Acids, Omega-3; Tears; Osmolar Concentration; Anterior Eye Segment; Severity of Illness Index
MeSH Terms: conditions — Dry Eye Syndromes; Lymphoma, Follicular; Lacerations

STUDY DESIGN:
Intervention Model Description: Part 1. Piiloset Trehalose Emulsion Eye Drop is administered on the worst eye four times during office hours of one day at the study centre.
  Part 2. Piiloset Trehalose Emulsion Eye Drop is self-administered on a randomized eye and the control eye drops on the contralateral eye three times a day for 10 days in a double-blinded fashion.
  Part 3. Either Piiloset Trehalose Emulsion Eye Drop or the control eye drops are self-administered on both eyes three times a day for 30 days in a randomized and double-blinded fashion.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emulsion Eye Drops (Experimental): Daily treatment with Piiloset Trehalose Emulsion Eye Drops
  Interventions: Device: Piiloset Trehalose Emulsion Eye Drops
- Control Eye Drops (Active Comparator): Daily treatment with Hyaluronic Acid Eye Drops (a CE-marked medical device)
  Interventions: Device: Control Eye Drops

INTERVENTIONS:
Device: Piiloset Trehalose Emulsion Eye Drops — Topical application of preservative-free multidose Piiloset Trehalose Emulsion Eye Drops 3 times daily
  Arms: Emulsion Eye Drops
Device: Control Eye Drops — Topical application of preservative-free multidose Hyaluronic Acid Eye Drops 3 times daily
  Arms: Control Eye Drops

SUMMARY:
The study evaluates the safety, ocular tolerability and efficacy of emulsion eye drops with sacha inchi seed oil, trehalose and hyaluronic acid in the treatment of moderate or severe dry eye in adult patients. The investigative device is studied in comparison with control eye drops containing hyaluronic acid for up to 30 days.

DETAILED DESCRIPTION:
According to the current view on dry eye disease, tear film instability, tear film hyperosmolarity, and ocular surface inflammation and damage are identified as etiological factors. The first-line medicinal management options include ocular lubricants such as eye drops and sprays. Emulsion eye drops are a relatively recent entity among topical therapies with an intention to account for deficiencies in the outermost lipid layer of the tear film.

Piiloset Trehalose Emulsion Eye Drops was developed to target and restore the three main layers (mucin, aqueous, and lipid) of the tear film and to counteract the key etiological factors leading to dry eye. Hyaluronic acid and the oil component are intended to restore tear film instability, the hypo-osmolar composition and trehalose as an osmoprotectant are intended to protect the ocular epithelium against hyperosmolarity, and ocular surface inflammation and cellular damage are prevented by the cytoprotective and/or anti-oxidative action of hyaluronic acid, trehalose, and sacha inchi oil components. Additional water binding in the tear film is provided by hyaluronic acid, trehalose, and glycerol. Lubricating the ocular surface by high-molecular-weight hyaluronic acid will extend the precorneal retention time. Adjustments made to certain physical and chemical parameters in the formulation are anticipated to improve tear film spreading and adhesion. The optically clear o/w emulsion formulation is free of preservatives, materials of animal origin, phosphates, or alcohol. The combined action of the individual components is expected to produce clinically relevant mitigation of the signs and symptoms of dry eye.

The study comprises three Parts with scheduled visits on Day 1 (all Parts) and on end-of-study date (Parts 2 and 3) to the study centre. Each study subject will participate in no more than one Part of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Ability and willingness to give informed written consent prior to any screening procedure after explanation of the nature and possible consequences of the study.
2. Age between 18 and 80 years.
3. At least two the following conditions (A and B):

   A. Symptomatic dry eye with OSDI score ≥20. AND B1. Tear film break-up time (TBUT) <10 seconds. OR B2. Positive ocular (corneal and conjunctival) staining pattern
4. Body weight at least 45 kg.
5. Under stable topical and/or systemic therapy for at least 4 weeks before the study procedures and apparent ability and willingness to abstain from other therapies until completion of the study period.
6. Ability and willingness to self-administer eye drops.
7. Ability and willingness to understand and fill in the OSDI questionnaire.
8. Ability and willingness to comply with the study protocol and other study-related procedures.

Exclusion Criteria:

1. History of ocular surgery, trauma, or refractive laser vision correction procedure less than 3 months earlier.
2. Evidence of acute or chronic infection in the cornea or conjunctiva.
3. Diagnosis of Sjögren's syndrome.
4. Unwillingness or apparent disability to discontinue contact lens use during study period and at least one week before the first dosing day.
5. Current ocular allergy symptoms.
6. Known allergy to any constituent of the trehalose emulsion eye drops or control eye drops.
7. Currently pregnant, nursing or planning to become pregnant before completion of the study period.
8. Any other condition that may, in the Investigator's opinion, jeopardize the safety or availability of the subject or adherence to the study protocol or may interfere with the interpretation of the results and would thus make the subject inappropriate for entry in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2018-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kai Kaarniranta, Professor, Principal Investigator — Kuopio University Hospital
Locations (1):
- Department of Ophthalmology, Kuopio University Hospital, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Laihia J, Jarvinen R, Wylegala E, Kaarniranta K. Disease aetiology-based design of multifunctional microemulsion eye drops for moderate or severe dry eye: a randomized, quadruple-masked and active-controlled clinical trial. Acta Ophthalmol. 2020 May;98(3):244-254. doi: 10.1111/aos.14252. Epub 2019 Oct 3. PMID 31579987

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study comprised three sequential parts. Parts 1 to 3 involved different participants each, thus no participant flow between parts (or periods) took place.
Units Other Than Participants: Eyes
Groups:
- Emulsion Eye Drops: Daily treatment with Piiloset Trehalose Emulsion Eye Drops
  Piiloset Trehalose Emulsion Eye Drops: Topical application of preservative-free multidose Piiloset Trehalose Emulsion Eye Drops
  * Part 1: on one eye 4 times during one day
  * Part 2: on one randomized eye 3 times a day for 10 days
  * Part 3: on both eyes 3 times a day for 30 days
- Control Eye Drops: Daily treatment with Hyaluronic Acid Eye Drops (a CE-marked medical device)
  Control Eye Drops: Topical application of preservative-free multidose Hyaluronic Acid Eye Drops
  * Part 1: not used
  * Part 2: on randomized contralateral eye 3 times a day for 10 days
  * Part 3: on both eyes 3 times a day for 30 days
Period: Part 1
Arm/Group | Emulsion Eye Drops | Control Eye Drops
Started | 3; 3 Eyes (Emulsion Eye Drops were used on one eye only.) | 0; 0 Eyes (Control Eye Drops were not used for Part 1.)
Completed | 3; 3 Eyes (No participant completing Part 1 was allowed to continue to Parts 2 or 3.) | 0; 0 Eyes
Not Completed | 0; 0 Eyes | 0; 0 Eyes
Period: Part 2
Arm/Group | Emulsion Eye Drops | Control Eye Drops
Started | 9; 9 Eyes (Emulsion Eye Drops were used on one randomized eye. Participants were different from Part 1.) | 9; 9 Eyes (Control Eye Drops were used on contralateral eye. Participants were different from Part 1.)
Completed | 9; 9 Eyes (No participant completing Part 2 was allowed to continue to Part 3.) | 9; 9 Eyes (No participant completing Part 2 was allowed to continue to Part 3.)
Not Completed | 0; 0 Eyes | 0; 0 Eyes
Period: Part 3
Arm/Group | Emulsion Eye Drops | Control Eye Drops
Started | 26; 0 Eyes (Emulsion Eye Drops were used on both eyes. Participants were different from Parts 1 and 2.) | 26; 0 Eyes (Control Eye Drops were used on both eyes. Participants were different from Parts 1 and 2.)
Completed | 24; 0 Eyes (Per-protocol (PP) dataset. 'Not Completed' participants are included in safety and ITT datasets.) | 25; 0 Eyes (Per-protocol (PP) dataset. 'Not Completed' participants are included in safety and ITT datasets.)
Not Completed | 2; 0 Eyes | 1; 0 Eyes
Not completed — Physician Decision | 1 | 0
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Population: Part 3: 52 eyes of 26 pts treated with Emulsion Eye Drops and 52 eyes of 26 pts treated with Control Eye Drops.
  Results are reported for Part 3 only.
Groups:
- Emulsion Eye Drops: Daily treatment with Piiloset Trehalose Emulsion Eye Drops
  Results are reported for Part 3 only:
  Topical application of preservative-free multidose Piiloset Trehalose Emulsion Eye Drops on both eyes 3 times a day for 30 days
- Control Eye Drops: Daily treatment with Hyaluronic Acid Eye Drops (a CE-marked medical device)
  Results are reported for Part 3 only:
  Topical application of preservative-free multidose Hyaluronic Acid Eye Drops on both eyes 3 times a day for 30 days
- Total: Total of all reporting groups
Arm/Group | Emulsion Eye Drops | Control Eye Drops | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (13.8) | 51.5 (11.4) | 53.3 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 8 | 8 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Finland | 26 | 26 | 52
Body Weight [Mean (Standard Deviation); unit: kg] | 75.1 (11.7) | 76.9 (15.8) | 76.0 (13.8)
Ocular Surface Disease Index (OSDI) [Mean (Standard Deviation); unit: units on a scale] — Ocular Surface Disease Index (OSDI) is a questionnaire consisting of 12 questions subdivided into 3 subscales for measuring the frequency of dry eye symptoms, vision-related quality of life and environmental triggers during the previous week. Answers to each question are on a scale of 0 (None of the time) to 4 (All of the time). Both total OSDI and its subscale scores are on a scale of 0 to 100, calculated as follows: score = (sum of scores for questions answered/number of questions answered) x 25. Higher scores represent greater disability.
  units on a scale | 48.1 (10.8) | 45.6 (11.3) | 46.9 (11.0)
Tear Break-Up Time (TBUT) [Mean (Standard Deviation); unit: s] | 3.35 (2.62) | 3.46 (2.04) | 3.40 (2.33)
Tear osmolarity [Mean (Standard Deviation); unit: mOsm/L] | 304.0 (11.8) | 307.3 (12.4) | 305.6 (12.1)
Blink rate [Mean (Standard Deviation); unit: Blinks/min] — Measurement of spontaneous eyelid blinks per minute
  Blinks/min | 18.17 (11.49) | 22.27 (12.93) | 20.22 (12.28)
Ocular protection index (OPI) [Mean (Standard Deviation); unit: ratio] — Ocular protection index (OPI) is the ratio of TBUT/IBI (IBI, interblink interval calculated from blink rate). An OPI value >1 indicates that TBUT (s) exceeds IBI (s) and that the ocular surface is mostly tear-film protected, because tear film break-ups do not take place within spontaneous blink cycles.
  ratio | 0.98 (0.937) | 1.23 (1.188) | 1.11 (1.067)
Corneal staining [Mean (Standard Deviation); unit: score on a scale] — Corneal staining score is assessed as the average number of punctate dots on an ordinal scale of 0, 1, 2, 3, 4, and 5 (Oxford scale) when compared to a pictorial standard. The number of dots increases on a log scale. Higher score represents more intense staining.
  score on a scale | 1.37 (0.794) | 1.21 (0.603) | 1.29 (0.703)
Conjunctival staining (temporal) [Mean (Standard Deviation); unit: score on a scale] — Conjunctival staining score is assessed as the average number of punctate dots on an ordinal scale of 0, 1, 2, 3, 4, and 5 (Oxford scale) when compared to a pictorial standard. The number of dots increases on a log scale. Higher score represents more intense staining.
  score on a scale | 1.06 (0.432) | 1.06 (0.497) | 1.06 (0.461)
Conjunctival staining (nasal) [Mean (Standard Deviation); unit: score on a scale] — Conjunctival staining score is assessed as the average number of punctate dots on an ordinal scale of 0, 1, 2, 3, 4, and 5 (Oxford scale) when compared to a pictorial standard. The number of dots increases on a log scale. Higher score represents more intense staining.
  score on a scale | 1.23 (0.430) | 1.23 (0.406) | 1.23 (0.414)
Conjunctival redness [Mean (Standard Deviation); unit: score on a scale] — Conjunctival redness score is assessed on an ordinal scale of 0 to 4 (Institute for Eye Research (IER) grading scale):
  0 = not existing, 1 = very slight, 2 = slight, 3 = moderate, 4 = severe. Higher score represents more intense redness.
  score on a scale | 1.98 (0.685) | 1.94 (0.829) | 1.96 (0.753)
Lid redness [Mean (Standard Deviation); unit: score on a scale] — Eyelid redness score is assessed on an ordinal scale of 0 to 4 (Institute for Eye Research (IER) grading scale):
  0 = not existing, 1 = very slight, 2 = slight, 3 = moderate, 4 = severe. Higher score represents more intense redness.
  score on a scale | 1.29 (0.751) | 1.29 (0.724) | 1.29 (0.730)
Intraocular pressure [Mean (Standard Deviation); unit: mmHg (Goldmann tonometer)] | 14.92 (2.134) | 15.69 (2.558) | 15.31 (2.364)
Ocular surgery, trauma, refractive laser vision correction [Count of Participants; unit: Participants] | 0 | 0 | 0
Eye infection [Count of Participants; unit: Participants] | 0 | 0 | 0
Allergy [Count of Participants; unit: Participants] | 0 | 0 | 0
Current or planned pregnancy and nursing [Count of Participants; unit: Participants] | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline OSDI
Description: Ocular Surface Disease Index (OSDI) is a questionnaire consisting of 12 questions subdivided into 3 subscales for measuring the frequency of dry eye symptoms, vision-related quality of life and environmental triggers during the previous week. Answers to each question are on a scale of 0 (None of the time) to 4 (All of the time). Both total OSDI and its subscale scores are on a scale of 0 to 100, calculated as follows: score = (sum of scores for questions answered/number of questions answered) x 25. Higher scores represent greater disability.
Time Frame: From baseline to Day 30 (Part 3)
Population: Intent-to-treat (ITT) dataset
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Emulsion Eye Drops | Control Eye Drops
Number analyzed (Participants) | 26 | 26
units on a scale | -24.64 (16.186) | -26.53 (14.620)
Statistical Analysis 1: Comparison: Emulsion Eye Drops vs Control Eye Drops; Between-group comparison, change from baseline; Test type: Superiority; p = 0.662, ANOVA — A two-sided p-value less than 0.05 was considered statistically significant; Mean Difference (Final Values) = 1.8837, 95% CI 2-sided [-6.7081 to 10.4756]
Statistical Analysis 2: Comparison: Emulsion Eye Drops; Within-group change from baseline; Test type: Other; p < 0.0001, ANOVA — A two-sided p-value less than 0.05 was considered statistically significant; Mean Difference (Final Values) = -24.6445, 95% CI 2-sided [-30.7199 to -18.5692]
Statistical Analysis 3: Comparison: Control Eye Drops; Within-group change from baseline; Test type: Other; p < 0.0001, ANOVA — A two-sided p-value less than 0.05 was considered statistically significant; Mean Difference (Final Values) = -26.5283, 95% CI 2-sided [-32.6036 to -20.4529]

2. Primary Outcome: Change From Baseline Tear Osmolarity
Description: Instrumental assay of tear fluid osmolarity (mOsm/L)
Time Frame: From baseline to Day 30 (Part 3)
Population: Intent-to-treat (ITT) dataset
Measure: Mean (Standard Deviation); unit: mOsm/L
Arm/Group | Emulsion Eye Drops | Control Eye Drops
Number analyzed (Participants) | 26 | 26
mOsm/L | -4.75 (16.224) | -1.77 (21.531)
Statistical Analysis 1: Comparison: Emulsion Eye Drops vs Control Eye Drops; Between-group comparison, change from baseline; Test type: Other; p = 0.575, ANOVA — A two-sided p-value less than 0.05 was considered statistically significant; Mean Difference (Final Values) = -2.9808, 95% CI 2-sided [-13.6005 to 7.6390]
Statistical Analysis 2: Comparison: Emulsion Eye Drops; Within-group change from baseline; Test type: Other; p = 0.2098, ANOVA — A two-sided p-value less than 0.05 was considered statistically significant; Mean Difference (Final Values) = -4.7500, 95% CI 2-sided [-12.2593 to 2.7593]
Statistical Analysis 3: Comparison: Control Eye Drops; Within-group change from baseline; Test type: Other; p = 0.6381, ANOVA — A two-sided p-value less than 0.05 was considered statistically significant; Mean Difference (Final Values) = -1.7692, 95% CI 2-sided [-9.2785 to 5.7401]

3. Primary Outcome: Change From Baseline TBUT
Description: Tear film break-up time (TBUT) (s)
Time Frame: From baseline to Day 30 (Part 3)
Population: Intent-to-treat (ITT) dataset
Measure: Mean (Standard Deviation); unit: s
Arm/Group | Emulsion Eye Drops | Control Eye Drops
Number analyzed (Participants) | 26 | 26
s | 1.71 (3.424) | 0.87 (1.809)
Statistical Analysis 1: Comparison: Emulsion Eye Drops vs Control Eye Drops; Between-group comparison, change from baseline; Test type: Other; p = 0.271, ANOVA — A two-sided p-value less than 0.05 was considered statistically significant; Mean Difference (Final Values) = 0.8462, 95% CI 2-sided [-0.6792 to 2.3715]
Statistical Analysis 2: Comparison: Emulsion Eye Drops; Within-group change from baseline; Test type: Other; p = 0.0025, ANOVA — A two-sided p-value less than 0.05 was considered statistically significant; Mean Difference (Final Values) = 1.7115, 95% CI 2-sided [0.6330 to 2.7901]
Statistical Analysis 3: Comparison: Control Eye Drops; Within-group change from baseline; Test type: Other; p = 0.1134, ANOVA — A two-sided p-value less than 0.05 was considered statistically significant; Mean Difference (Final Values) = 0.8654, 95% CI 2-sided [-0.2132 to 1.9440]

4. Secondary Outcome: Change From Baseline Blink Rate
Description: Measurement of spontaneous eyelid blinks per minute
Time Frame: From baseline to Day 30 (Part 3)
Population: Intent-to-treat (ITT) dataset
Measure: Mean (Standard Deviation); unit: Blinks/min
Arm/Group | Emulsion Eye Drops | Control Eye Drops
Number analyzed (Participants) | 26 | 26
Blinks/min | 0.02 (8.721) | -2.15 (10.161)
Statistical Analysis 1: Comparison: Emulsion Eye Drops vs Control Eye Drops; Between-group comparison, change from baseline; Test type: Other; p = 0.412, ANOVA — A two-sided p-value less than 0.05 was considered statistically significant; Mean Difference (Final Values) = 2.1731, 95% CI 2-sided [-3.1016 to 7.4477]
Statistical Analysis 2: Comparison: Emulsion Eye Drops; Within-group change from baseline; Test type: Other; p = 0.9918, ANOVA — A two-sided p-value less than 0.05 was considered statistically significant; Mean Difference (Final Values) = 0.01923, 95% CI 2-sided [-3.7105 to 3.7490]
Statistical Analysis 3: Comparison: Control Eye Drops; Within-group change from baseline; Test type: Other; p = 0.2516, ANOVA — A two-sided p-value less than 0.05 was considered statistically significant; Mean Difference (Final Values) = -2.1538, 95% CI 2-sided [-5.8836 to 1.5759]

5. Secondary Outcome: Change From Baseline Ocular Protection Index (OPI)
Description: OPI is the ratio of TBUT/IBI (IBI, interblink interval calculated from blink rate). An OPI value >1 indicates that TBUT (s) exceeds IBI (s) and that the ocular surface is mostly tear-film protected, because tear film break-ups do not take place within spontaneous blink cycles.
Time Frame: From baseline to Day 30 (Part 3)
Population: Intent-to-treat (ITT) dataset
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Emulsion Eye Drops | Control Eye Drops
Number analyzed (Participants) | 26 | 26
ratio | 0.56 (1.078) | 0.05 (0.680)
Statistical Analysis 1: Comparison: Emulsion Eye Drops vs Control Eye Drops; Between-group comparison, change from baseline; Test type: Other; p = 0.047, ANOVA — A two-sided p-value less than 0.05 was considered statistically significant; Mean Difference (Final Values) = 0.5093, 95% CI 2-sided [0.007267 to 1.0113]
Statistical Analysis 2: Comparison: Emulsion Eye Drops; Within-group change from baseline; Test type: Other; p = 0.0026, ANOVA — A two-sided p-value less than 0.05 was considered statistically significant; Mean Difference (Final Values) = 0.5596, 95% CI 2-sided [0.2046 to 0.9146]
Statistical Analysis 3: Comparison: Control Eye Drops; Within-group change from baseline; Test type: Other; p = 0.7770, ANOVA — A two-sided p-value less than 0.05 was considered statistically significant; Mean Difference (Final Values) = 0.05032, 95% CI 2-sided [-0.3047 to 0.4053]

6. Secondary Outcome: Change From Baseline Corneal Staining
Description: Corneal staining score is assessed as the average number of punctate dots on an ordinal scale of 0, 1, 2, 3, 4, and 5 (Oxford scale) when compared to a pictorial standard. The number of dots increases on a log scale. Higher score represents more intense staining.
Time Frame: From baseline to Day 30 (Part 3)
Population: Per-protocol (PP) dataset
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Emulsion Eye Drops | Control Eye Drops
Number analyzed (Participants) | 24 | 25
score on a scale | -0.38 (0.695) | -0.22 (0.522)
Statistical Analysis 1: Comparison: Emulsion Eye Drops vs Control Eye Drops; Between-group comparison, change from baseline; Test type: Other; p = 0.447, Wilcoxon rank sum test — A two-sided p-value less than 0.05 was considered statistically significant; Wilcoxon Z statistic = -0.7604
Statistical Analysis 2: Comparison: Emulsion Eye Drops; Within-group change from baseline; Test type: Other; p = 0.014, Wilcoxon rank sum test — A two-sided p-value less than 0.05 was considered statistically significant
Statistical Analysis 3: Comparison: Control Eye Drops; Within-group change from baseline; Test type: Other; p = 0.070, Wilcoxon rank sum test — A two-sided p-value less than 0.05 was considered statistically significant

7. Secondary Outcome: Change From Baseline Conjunctival (Temporal) Staining
Description: Conjunctival staining score is assessed as the average number of punctate dots on an ordinal scale of 0, 1, 2, 3, 4, and 5 (Oxford scale) when compared to a pictorial standard. The number of dots increases on a log scale. Higher score represents more intense staining.
Time Frame: From baseline to Day 30 (Part 3)
Population: Per-protocol (PP) dataset
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Emulsion Eye Drops | Control Eye Drops
Number analyzed (Participants) | 24 | 25
score on a scale | -0.19 (0.507) | -0.02 (0.810)
Statistical Analysis 1: Comparison: Emulsion Eye Drops vs Control Eye Drops; Between-group comparison, change from baseline; Test type: Other; p = 0.522, Wilcoxon rank sum test — A two-sided p-value less than 0.05 was considered statistically significant; Wilcoxon Z statistic = -0.6396
Statistical Analysis 2: Comparison: Emulsion Eye Drops; Within-group change from baseline; Test type: Other; p = 0.119, Wilcoxon rank sum test — A two-sided p-value less than 0.05 was considered statistically significant
Statistical Analysis 3: Comparison: Control Eye Drops; Within-group change from baseline; Test type: Other; p = 0.900, Wilcoxon rank sum test — A two-sided p-value less than 0.05 was considered statistically significant

8. Secondary Outcome: Change From Baseline Conjunctival (Nasal) Staining
Description: as for outcome 7
Time Frame: From baseline to Day 30 (Part 3)
Population: Per-protocol (PP) dataset
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Emulsion Eye Drops | Control Eye Drops
Number analyzed (Participants) | 24 | 25
score on a scale | -0.27 (0.608) | -0.12 (0.666)
Statistical Analysis 1: Comparison: Emulsion Eye Drops vs Control Eye Drops; Between-group comparison, change from baseline; Test type: Other; p = 0.590, Wilcoxon rank sum test — A two-sided p-value less than 0.05 was considered statistically significant; Wilcoxon Z statistic = -0.5387
Statistical Analysis 2: Comparison: Emulsion Eye Drops; Within-group change from baseline; Test type: Other; p = 0.043, Wilcoxon rank sum test — A two-sided p-value less than 0.05 was considered statistically significant
Statistical Analysis 3: Comparison: Control Eye Drops; Within-group change from baseline; Test type: Other; p = 0.442, Wilcoxon rank sum test — A two-sided p-value less than 0.05 was considered statistically significant

9. Other Pre Specified Outcome: Change From Baseline Visual Acuity
Description: Best corrected visual acuity (ETDRS charts 1 & 2, 2000 series)
Time Frame: From baseline to Day 30 (Part 3)
Population: Safety dataset
Measure: Mean (Standard Deviation); unit: logMAR chart log units
Arm/Group | Emulsion Eye Drops | Control Eye Drops
Number analyzed (Participants) | 26 | 26
logMAR chart log units | -0.03 (0.071) | -0.04 (0.080)

10. Other Pre Specified Outcome: Change From Baseline Conjunctival Redness
Description: Conjunctival redness score is assessed on an ordinal scale of 0 to 4 (IER grading scale):
  0 = not existing, 1 = very slight, 2 = slight, 3 = moderate, 4 = severe. Higher score represents more intense redness.
Time Frame: From baseline to Day 30 (Part 3)
Population: Safety dataset
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Emulsion Eye Drops | Control Eye Drops
Number analyzed (Participants) | 26 | 26
score on a scale | -0.46 (0.647) | -0.27 (0.652)
Statistical Analysis 1: Comparison: Emulsion Eye Drops vs Control Eye Drops; Between-group comparison, change from baseline; Test type: Other; p = 0.357, Wilcoxon rank sum test — A two-sided p-value less than 0.05 was considered statistically significant; Wilcoxon Z statistic = 0.9208
Statistical Analysis 2: Comparison: Emulsion Eye Drops; Within-group change from baseline; Test type: Other; p = 0.001, Wilcoxon rank sum test — A two-sided p-value less than 0.05 was considered statistically significant
Statistical Analysis 3: Comparison: Control Eye Drops; Within-group change from baseline; Test type: Other; p = 0.065, Wilcoxon rank sum test — A two-sided p-value less than 0.05 was considered statistically significant

11. Other Pre Specified Outcome: Change From Baseline Lid Redness
Description: Eyelid redness score is assessed on an ordinal scale of 0 to 4 (IER grading scale):
  0 = not existing, 1 = very slight, 2 = slight, 3 = moderate, 4 = severe. Higher score represents more intense redness.
Time Frame: From baseline to Day 30 (Part 3)
Population: Safety dataset
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Emulsion Eye Drops | Control Eye Drops
Number analyzed (Participants) | 26 | 26
score on a scale | -0.37 (0.672) | -0.19 (0.549)
Statistical Analysis 1: Comparison: Emulsion Eye Drops vs Control Eye Drops; Between-group comparison, change from baseline; Test type: Other; p = 0.296, Wilcoxon rank sum test — A two-sided p-value less than 0.05 was considered statistically significant; Wilcoxon Z statistic = 1.0440
Statistical Analysis 2: Comparison: Emulsion Eye Drops; Within-group change from baseline; Test type: Other; p = 0.012, Wilcoxon rank sum test — A two-sided p-value less than 0.05 was considered statistically significant
Statistical Analysis 3: Comparison: Control Eye Drops; Within-group change from baseline; Test type: Other; p > 0.05, Wilcoxon rank sum test — A two-sided p-value less than 0.05 was considered statistically significant

12. Other Pre Specified Outcome: Change From Baseline Intraocular Pressure
Description: Intraocular pressure measured using Goldmann applanation tonometry (mmHg)
Time Frame: From baseline to Day 30 (Part 3)
Population: Safety dataset
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Emulsion Eye Drops | Control Eye Drops
Number analyzed (Participants) | 26 | 26
mmHg | -0.12 (1.705) | -0.42 (1.653)

13. Post Hoc Outcome: Change From Baseline Tear Osmolarity in Hyperosmolar Participants
Description: Instrumental assay of tear fluid osmolarity (mOsm/L) in a hyperosmolar subgroup of participants (mean of eyes ≥308 mOsm/L)
Time Frame: From baseline to Day 30 (Part 3)
Population: ITT population with hyperosmolar tears (mean of eyes ≥308 mOsm/L)
Measure: Mean (Standard Deviation); unit: mOsm/L
Arm/Group | Emulsion Eye Drops | Control Eye Drops
Number analyzed (Participants) | 8 | 14
mOsm/L | -17.06 (10.425) | -15.07 (16.596)
Statistical Analysis 1: Comparison: Emulsion Eye Drops vs Control Eye Drops; Between-group comparison, change from baseline; Test type: Other; p = 0.764, ANOVA — A two-sided p-value less than 0.05 was considered statistically significant; Mean Difference (Final Values) = -1.9911, 95% CI 2-sided [-15.6117 to 11.6295]
Statistical Analysis 2: Comparison: Emulsion Eye Drops; Within-group change from baseline; Test type: Other; p = 0.0038, ANOVA — A two-sided p-value less than 0.05 was considered statistically significant; Mean Difference (Final Values) = -17.0625, 95% CI 2-sided [-27.9280 to -6.1970]
Statistical Analysis 3: Comparison: Control Eye Drops; Within-group change from baseline; Test type: Other; p = 0.0011, ANOVA — A two-sided p-value less than 0.05 was considered statistically significant; Mean Difference (Final Values) = -15.0714, 95% CI 2-sided [-23.2850 to -6.8579]

ADVERSE EVENTS:
Time Frame: Part 1: 1 day; Part 2: 10 days; Part 3: 30 days
Description: ADE (adverse device effect); AE (adverse event); SADE (serious adverse device effect); SAE (serious adverse event); USADE (unanticipated serious adverse device effect)
  Total Number of Participants at Risk (safety population); Emulsion Eye Drops: 3 + 9 + 26 = 38 participants; Control Eye Drops: 0 + 9 + 26 = 35 participants.
  Adverse events were collected throughout the study during visits to study site, in study diaries, and from direct contacts to study personnel between visits.
Groups:
- Emulsion Eye Drops: Daily treatment with Piiloset Trehalose Emulsion Eye Drops
  Adverse events are reported for the safety population in all parts of the study, including all randomized subjects who received Piiloset Trehalose Emulsion Eye Drops at least once and from whom at least one safety measurement was obtained after randomization.
- Control Eye Drops: Daily treatment with Hyaluronic Acid Eye Drops (a CE-marked medical device)
  Adverse events are reported for the safety population in all parts of the study, including all randomized subjects who received Hyaluronic Acid Eye Drops at least once and from whom at least one safety measurement was obtained after randomization.
Arm/Group | Emulsion Eye Drops | Control Eye Drops
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/35
Other Adverse Events (participants affected / at risk) | 1/38 | 0/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emulsion Eye Drops (N=38) | Control Eye Drops (N=35)
AE (adverse event) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Small cutaneous papules all over the body, judged by the Investigator to be unrelated to study treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restrictions on the PI are that the sponsor can review results communications 30 days prior to planned date of public release. If public release of information in communications may jeopardize protecting sponsor's immaterial rights, the sponsor can additionally embargo the communications for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2018-04-06): https://cdn.clinicaltrials.gov/large-docs/02/NCT03569202/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-06): https://cdn.clinicaltrials.gov/large-docs/02/NCT03569202/SAP_001.pdf